CLINICAL TRIAL: NCT01455597
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of WC3011 (Estradiol Vaginal Cream) in the Treatment of Symptoms of Vulvovaginal Atrophy in Postmenopausal Women
Brief Title: Evaluate Long-Term Safety and Efficacy WC3011 (Estradiol Vaginal Cream)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-04509
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-09

CONDITIONS: Vulvovaginal Atrophy
Keywords: Postmenopausal Women; Vaginal Dryness; Postmenopausal Vulvovaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WC3011 Estradiol Vaginal Cream (Experimental): WC3011 estradiol vaginal cream 3 times a week for up to 40 weeks.
  Interventions: Drug: WC3011 Estradiol Vaginal Cream

INTERVENTIONS:
Drug: WC3011 Estradiol Vaginal Cream — WC3011 estradiol vaginal cream, 3 times a week for 40 weeks.

SUMMARY:
This is an open-label extension study evaluating the long-term safety and efficacy of WC3011 in non-hysterectomized, healthy, postmenopausal women with vulvovaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study PR-04409.3 (NCT01400776)

Exclusion Criteria:

Developed any of the following during Study-PR04409.3 or has begun taking hormone therapy other than WC3011:

* Hypersensitivity to estrogen and/or progestin therapy
* Known or suspected premalignant or malignant disease (except successfully treated skin cancers)
* Manifestation of or treatment for significant cardiovascular disease, stroke or ischemic attack
* Insulin-dependent diabetes mellitus
* Smoking ≥ 15 cigarettes daily
* Uncontrolled hypertension - systolic blood pressure (BP) ≥ 160 mmHG or diastolic ≥ 95 mmHg

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was to treat the symptoms of vulvovaginal atrophy in postmenopausal women.
Enrollment: 309 (Actual)
Dates: Start 2011-10-20 (Actual); Primary Completion 2012-12-03 (Actual); Study Completion 2012-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, PharmD, Study Director — Allergan
Locations (64):
- United States (64):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Warner Chilcott Investigational Site, Mobile, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials, LLC, Phoenix, Arizona
  - Radiant Research-Scottsdale, Scottsdale, Arizona
  - Radiant Research-Tucson, Tucson, Arizona
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Healthcare Inc., San Diego, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - New Age Medical Research Corp, Miami, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - OB-GYN Specialists of the Palm Beaches, Palm Beach Gardens, Florida
  - Radiant Research-St. Petersburg, Pinellas Park, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Radiant Research-Atlanta, Atlanta, Georgia
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - Radiant Research-Chicago, Chicago, Illinois
  - Springfield Clinical, LLP, Springfield, Illinois
  - The South Bend Clinic, LLP, Granger, Indiana
  - Radiant Research - Overland Park, Overland Park, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - York Clinical Consulting, Marrero, Louisiana
  - Women Under Study, New Orleans, Louisiana
  - Beyer Research, Kalamazoo, Michigan
  - Ridgeview Research, Chaska, Minnesota
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Office of R. Garn Mabey, M.D., Las Vegas, Nevada
  - Lawrence OB-GYN Associates, P.C., Lawrenceville, New Jersey
  - Phoenix OB-GYN Assoc., LLC, Moorestown, New Jersey
  - Women's Health Research Center, Plainsboro, New Jersey
  - Hawthorne Medical Research, Inc., Greensboro, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - The Columbus Center for Women's Health Research, Columbus, Ohio
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Advanced Clinical Research, Medford, Oregon
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Susan L. Floyd, MD, PC, Wexford, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Fellows Research Alliance, Inc., Bluffton, South Carolina
  - Practice Research Organization, Inc., Dallas, Texas
  - Radiant Research-Dallas, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Advances In Health, Inc, Houston, Texas
  - Radiant Research-San Antonio, San Antonio, Texas
  - Center for Reproductive Medicine, Webster, Texas
  - J. Lewis Research-Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research - Foothill Family Clinic South, Salt Lake City, Utah
  - Physicians' Research Options LLC, Sandy City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Women's Center, Richmond, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - North Spokane Women's Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed study PR-04409.3 (NCT01400776) were enrolled to receive W13011 estradiol vaginal cream three times a week in this study. Participant flow and outcome measures data were summarized as per treatment received in previous study.
Groups:
- Previous WC3011 Estradiol Vaginal Cream (2 Times/Week): WC3011 estradiol vaginal cream. applied vaginally 3 times a week for up to 40 weeks in this study (Participants who received WC3011 estradiol vaginal cream 2 times a week in the previous study were included in this arm group).
- Previous Vehicle (2 Times/Week): WC3011 estradiol vaginal cream applied vaginally 3 times a week for up to 40 weeks in this study (Participants who received vehicle 2 times a week in the previous study were included in this arm group).
- Previous WC3011 Estradiol Vaginal Cream (3 Times/Week): WC3011 estradiol vaginal cream applied vaginally 3 times a week for up to 40 weeks in this study (Participants who received WC13011 estradiol vaginal cream 3 times a week in the previous study were included in this arm group).
- Previous Vehicle (3 Times/Week): WC3011 estradiol vaginal cream applied vaginally 3 times a week for up to 40 weeks in this study (Participants who received vehicle 3 times a week in the previous study were included in this arm group).
Period: Overall Study
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Started | 101 | 56 | 100 | 52
All-Participants-Treated Population (All enrolled participants who received at least 1 dose of study drug in Study PR-04509.) | 101 | 56 | 99 | 52
Completed | 84 | 48 | 80 | 42
Not Completed | 17 | 8 | 20 | 10
Not completed — Adverse Event | 7 | 0 | 5 | 1
Not completed — Lack of Efficacy | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1
Not completed — Withdrew Consent | 6 | 5 | 8 | 5
Not completed — Reason not Specified | 1 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug in Study PR-04509.
Groups:
- WC3011 Estradiol Vaginal Cream: WC3011 estradiol vaginal cream applied vaginally 3 times a week for up to 40 weeks.
Arm/Group | WC3011 Estradiol Vaginal Cream
Number analyzed (Participants) | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Endometrial Biopsy Results at Final Visit
Description: The endometrial biopsy results was categorized as: normal results categorized as atrophic/inactive or proliferative, unsatisfactory with endometrial thickness ≤4 mm and missing biopsy with endometrial thickness ≤4 mm; abnormal results categorized as polyp, hyperplasia, and carcinoma; unknown result categorized as unsatisfactory with endometrial thickness >4 mm, missing biopsy with endometrial thickness >4 mm, unsatisfactory without transvaginal ultrasonography (TVU) result and missing biopsy without TVU result. The duration of estradiol exposure was combination of studies PR-04409.3 and PR-04509.
Time Frame: Final Visit (Day closest to Day 281)
Population: All participants who received at least 1 dose of study drug in Study PR-04509. Data is reported as per the duration of exposure of participants receiving study treatment. Overall number analyzed is the number of participants with available data at the given timepoint. Only categories for which there was at least 1 participant are reported.
Measure: Count of Participants; unit: Participants
Groups:
- WC3011 Estradiol Vaginal Cream: Less Than 92 Days: WC3011 estradiol vaginal cream applied vaginally 3 times a week for a median exposure of less than 92 days.
- WC3011 Estradiol Vaginal Cream: 92-182 Days: WC3011 estradiol vaginal cream applied vaginally 3 times a week for median exposure of 92 to 182 days.
- WC3011 Estradiol Vaginal Cream: 183-273 Days: WC3011 estradiol vaginal cream applied vaginally 3 times a week for median exposure of 183 to 273 days.
- WC3011 Estradiol Vaginal Cream: More Than 273 Days: WC3011 estradiol vaginal cream applied vaginally 3 times a week for median exposure of more than 273 days.
Arm/Group | WC3011 Estradiol Vaginal Cream: Less Than 92 Days | WC3011 Estradiol Vaginal Cream: 92-182 Days | WC3011 Estradiol Vaginal Cream: 183-273 Days | WC3011 Estradiol Vaginal Cream: More Than 273 Days
Number analyzed (Participants) | 7 | 27 | 19 | 255
Participants
  Normal Biopsy: Atrophic | 3 | 10 | 7 | 166
  Normal Biopsy: Proliferative | 0 | 1 | 1 | 3
  Normal Biopsy: Unsatisfactory With Endometrial Thickness ≤4 mm | 0 | 3 | 4 | 48
  Normal Biopsy: Missing Biopsy With Endometrial Thickness ≤4 mm | 1 | 1 | 1 | 21
  Abnormal Biopsy: Polyp | 0 | 0 | 0 | 1
  Unknown: Unsatisfactory With Endometrial Thickness >4 mm | 0 | 1 | 0 | 6
  Unknown: Missing Biopsy With Endometrial Thickness >4 mm | 0 | 0 | 0 | 1
  Unknown: Unsatisfactory Without TVU Result | 0 | 2 | 0 | 3
  Unknown: Missing Biopsy Without TVU Result | 3 | 9 | 6 | 6

2. Secondary Outcome: Change From Baseline in Participants Self-Assessment of the Symptoms of Vulvovaginal Atrophy (VVA) at Each Post-baseline Timepoints
Description: Self-Assessment of the symptoms of VVA was evaluated for vaginal dryness, vaginal Itching, dysuria, and dyspareunia by a questionnaire. Questionnaire consisted of 5 questions scaled from 0 to 3 level of intensity, where 0-none indicated symptom not present; 1-mild indicated symptom is present but may be intermittent; does not interfere with your activities or lifestyle; 2-moderate indicated symptom is present, aware of the symptom but activities and lifestyle are only occasionally affected; 3-severe indicated usually aware and bothered by the symptom and have modified your activities and/or lifestyle due to the symptom. Higher score indicated most bothersome symptoms. A negative change from Baseline indicates improvement. Participants at Final visit/Visit 7 included those who were to complete all the evaluations in the study including who prematurely withdrew from the study.
Time Frame: Baseline (Baseline/Visit 1 for this study was the same as Final Visit/Visit 5 for completers of PR-04409.3) to Weeks 4, 8, 16, 24, 32, 40 and Final Visit (Day closest to Day 281)
Population: All participants who received at least 1 dose of study drug in Study PR-04509. Number analyzed is the number of participants with available data at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Number analyzed (Participants) | 101 | 56 | 99 | 52
score on a scale
  Vaginal Dryness-Baseline | 1.2 (0.92) | 1.5 (0.91) | 1.2 (0.87) | 1.5 (1.06)
  Vaginal Dryness-Change From Baseline to Week 4: number analyzed (Participants) | 101 | 56 | 96 | 52
  Vaginal Dryness-Change From Baseline to Week 4 | -0.3 (0.71) | -0.3 (0.79) | -0.3 (0.62) | -0.2 (0.61)
  Vaginal Dryness-Change From Baseline to Week 8: number analyzed (Participants) | 100 | 53 | 96 | 51
  Vaginal Dryness-Change From Baseline to Week 8 | -0.4 (0.81) | -0.5 (0.80) | -0.4 (0.65) | -0.4 (0.64)
  Vaginal Dryness-Change From Baseline to Week 16: number analyzed (Participants) | 92 | 53 | 92 | 48
  Vaginal Dryness-Change From Baseline to Week 16 | -0.5 (0.75) | -0.6 (0.91) | -0.4 (0.72) | -0.3 (0.80)
  Vaginal Dryness-Change From Baseline to Week 24: number analyzed (Participants) | 90 | 50 | 89 | 43
  Vaginal Dryness-Change From Baseline to Week 24 | -0.6 (0.80) | -0.6 (0.78) | -0.3 (0.72) | -0.3 (0.85)
  Vaginal Dryness-Change From Baseline to Week 32: number analyzed (Participants) | 86 | 49 | 83 | 43
  Vaginal Dryness-Change From Baseline to Week 32 | -0.5 (0.88) | -0.7 (0.75) | -0.3 (0.68) | -0.4 (0.95)
  Vaginal Dryness-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Vaginal Dryness-Change From Baseline to Week 40 | -0.5 (0.87) | -0.6 (0.86) | -0.4 (0.78) | -0.5 (0.94)
  Vaginal Dryness-Change From Baseline to Final Visit: number analyzed (Participants) | 101 | 56 | 97 | 52
  Vaginal Dryness-Change From Baseline to Final Visit | -0.4 (0.89) | -0.6 (0.89) | -0.3 (0.76) | -0.5 (0.90)
  Vaginal Itching-Baseline | 0.6 (0.73) | 0.5 (0.71) | 0.5 (0.70) | 0.5 (0.67)
  Vaginal Itching-Change From Baseline to Week 4: number analyzed (Participants) | 101 | 56 | 96 | 52
  Vaginal Itching-Change From Baseline to Week 4 | -0.3 (0.63) | -0.0 (0.66) | -0.2 (0.60) | -0.0 (0.80)
  Vaginal Itching-Change From Baseline to Week 8: number analyzed (Participants) | 100 | 53 | 96 | 51
  Vaginal Itching-Change From Baseline to Week 8 | -0.2 (0.74) | -0.1 (0.64) | -0.3 (0.63) | 0.0 (0.68)
  Vaginal Itching-Change From Baseline to Week 16: number analyzed (Participants) | 92 | 53 | 92 | 48
  Vaginal Itching-Change From Baseline to Week 16 | -0.3 (0.77) | -0.0 (0.69) | -0.1 (0.70) | 0.1 (0.47)
  Vaginal Itching-Change From Baseline to Week 24: number analyzed (Participants) | 90 | 50 | 89 | 43
  Vaginal Itching-Change From Baseline to Week 24 | -0.3 (0.74) | -0.2 (0.59) | -0.2 (0.72) | 0.0 (0.58)
  Vaginal Itching-Change From Baseline to Week 32: number analyzed (Participants) | 86 | 49 | 83 | 43
  Vaginal Itching-Change From Baseline to Week 32 | -0.2 (0.69) | -0.2 (0.64) | -0.2 (0.64) | -0.1 (0.59)
  Vaginal Itching-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Vaginal Itching-Change From Baseline to Week 40 | -0.3 (0.80) | -0.3 (0.66) | -0.3 (0.71) | -0.0 (0.47)
  Vaginal Itching-Change From Baseline to Final Visit: number analyzed (Participants) | 101 | 56 | 97 | 52
  Vaginal Itching-Change From Baseline to Final Visit | -0.3 (0.78) | -0.3 (0.67) | -0.3 (0.71) | -0.0 (0.64)
  Dysuria-Baseline | 0.1 (0.42) | 0.2 (0.49) | 0.1 (0.33) | 0.1 (0.43)
  Dysuria-Change From Baseline to Week 4: number analyzed (Participants) | 101 | 56 | 96 | 52
  Dysuria-Change From Baseline to Week 4 | -0.1 (0.37) | -0.0 (0.50) | -0.0 (0.25) | -0.1 (0.33)
  Dysuria-Change From Baseline to Week 8: number analyzed (Participants) | 100 | 53 | 96 | 51
  Dysuria-Change From Baseline to Week 8 | -0.1 (0.41) | -0.0 (0.44) | 0.0 (0.35) | -0.0 (0.20)
  Dysuria-Change From Baseline to Week 16: number analyzed (Participants) | 92 | 53 | 92 | 48
  Dysuria-Change From Baseline to Week 16 | -0.1 (0.41) | -0.1 (0.51) | -0.0 (0.28) | 0.0 (0.14)
  Dysuria-Change From Baseline to Week 24: number analyzed (Participants) | 90 | 50 | 89 | 43
  Dysuria-Change From Baseline to Week 24 | -0.1 (0.29) | -0.2 (0.47) | -0.0 (0.28) | 0.0 (0.21)
  Dysuria-Change From Baseline to Week 32: number analyzed (Participants) | 86 | 49 | 83 | 43
  Dysuria-Change From Baseline to Week 32 | -0.1 (0.33) | -0.1 (0.54) | -0.0 (0.29) | 0.0 (0.22)
  Dysuria-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Dysuria-Change From Baseline to Week 40 | -0.1 (0.30) | -0.1 (0.41) | 0.0 (0.37) | 0.0 (0.27)
  Dysuria-Change From Baseline to Final Visit: number analyzed (Participants) | 101 | 56 | 97 | 52
  Dysuria-Change From Baseline to Final Visit | -0.1 (0.32) | -0.1 (0.49) | 0.0 (0.40) | 0.0 (0.28)
  Dyspareunia-Baseline: number analyzed (Participants) | 88 | 53 | 89 | 49
  Dyspareunia-Baseline | 1.3 (1.14) | 1.3 (1.14) | 1.2 (1.08) | 1.6 (1.24)
  Dyspareunia-Change From Baseline to Week 4: number analyzed (Participants) | 65 | 46 | 62 | 38
  Dyspareunia-Change From Baseline to Week 4 | -0.3 (0.69) | -0.5 (0.69) | -0.2 (0.66) | -0.5 (0.80)
  Dyspareunia-Change From Baseline to Week 8: number analyzed (Participants) | 66 | 42 | 62 | 40
  Dyspareunia-Change From Baseline to Week 8 | -0.3 (0.82) | -0.5 (0.77) | -0.3 (0.63) | -0.5 (1.13)
  Dyspareunia-Change From Baseline to Week 16: number analyzed (Participants) | 57 | 44 | 67 | 36
  Dyspareunia-Change From Baseline to Week 16 | -0.5 (0.93) | -0.6 (0.85) | -0.4 (0.83) | -0.5 (0.88)
  Dyspareunia-Change From Baseline to Week 24: number analyzed (Participants) | 57 | 43 | 62 | 30
  Dyspareunia-Change From Baseline to Week 24 | -0.6 (0.96) | -0.6 (0.85) | -0.4 (0.86) | -0.6 (1.01)
  Dyspareunia-Change From Baseline to Week 32: number analyzed (Participants) | 57 | 42 | 59 | 30
  Dyspareunia-Change From Baseline to Week 32 | -0.5 (0.95) | -0.7 (0.94) | -0.4 (0.78) | -0.6 (0.93)
  Dyspareunia-Change From Baseline to Week 40: number analyzed (Participants) | 56 | 39 | 61 | 30
  Dyspareunia-Change From Baseline to Week 40 | -0.6 (0.99) | -0.5 (0.82) | -0.3 (0.72) | -0.7 (1.06)
  Dyspareunia-Change From Baseline to Final Visit: number analyzed (Participants) | 74 | 50 | 78 | 42
  Dyspareunia-Change From Baseline to Final Visit | -0.5 (0.94) | -0.6 (0.91) | -0.3 (0.72) | -0.6 (1.15)

3. Secondary Outcome: Change From Baseline in Vaginal Cytology: Percentage of Superficial Vaginal Cells
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of superficial cells. Participants at Final visit/Visit 7 included those who were to complete all the evaluations in the study including who prematurely withdrew from the study.
Time Frame: Baseline (Baseline/Visit 1 for this study was the same as Final Visit/Visit 5 for completers of PR-04409.3) to Week 40 and Final Visit (Day closest to Day 281)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of superficial cells
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Number analyzed (Participants) | 101 | 56 | 99 | 52
percentage of superficial cells
  Baseline | 10.4 (11.73) | 4.0 (7.72) | 16.1 (18.77) | 3.1 (7.99)
  Change From Baseline to Week 40: number analyzed (Participants) | 69 | 40 | 73 | 35
  Change From Baseline to Week 40 | 12.8 (21.26) | 17.6 (18.21) | 0.5 (20.69) | 13.9 (24.56)
  Change From Baseline to Final Visit: number analyzed (Participants) | 85 | 48 | 85 | 41
  Change From Baseline to Final Visit | 11.0 (20.98) | 15.9 (17.59) | -0.2 (21.79) | 13.0 (23.02)

4. Secondary Outcome: Change From Baseline in Vaginal Cytology: Percentage of Parabasal Vaginal Cells
Description: Vaginal wall smears were collected from each participant. The smears were sent to the central laboratory for analysis to determine the percentage of parabasal cells. Participants at Final visit/Visit 7 included those who were to complete all the evaluations in the study including who prematurely withdrew from the study.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of parabasal cells
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Number analyzed (Participants) | 101 | 56 | 99 | 52
percentage of parabasal cells
  Baseline | 9.7 (24.34) | 42.2 (41.46) | 12.0 (29.28) | 34.2 (38.74)
  Change From Baseline to Week 40: number analyzed (Participants) | 69 | 40 | 73 | 35
  Change From Baseline to Week 40 | 0.0 (20.78) | -42.2 (42.00) | -1.5 (33.28) | -21.2 (36.83)
  Change From Baseline to Final Visit: number analyzed (Participants) | 85 | 48 | 85 | 41
  Change From Baseline to Final Visit | -0.4 (22.30) | -36.3 (43.18) | 1.2 (34.67) | -24.0 (36.80)

5. Secondary Outcome: Change From Baseline in Vaginal pH
Description: Vaginal pH was obtained at final visit of the study. The pH was a numeric value from 0 to 14 expressing the acidity or alkalinity of the vaginal fluids where 7 was neutral, lower values were more acidic (values of 0-6) and higher values more alkaline (values of 8-14). A negative change from Baseline indicates improvement. Participants at Final visit/Visit 7 included those who were to complete all the evaluations in the study including who prematurely withdrew from the study.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Number analyzed (Participants) | 101 | 56 | 99 | 52
score on a scale
  Baseline | 5.5 (0.81) | 6.2 (1.06) | 5.4 (0.80) | 6.1 (0.99)
  Change From Baseline to Week 40: number analyzed (Participants) | 83 | 48 | 80 | 42
  Change From Baseline to Week 40 | -0.3 (0.97) | -1.0 (1.24) | -0.2 (1.04) | -0.8 (0.95)
  Change From Baseline to Final Visit: number analyzed (Participants) | 95 | 54 | 93 | 49
  Change From Baseline to Final Visit | -0.2 (1.04) | -1.0 (1.19) | -0.1 (1.08) | -1.0 (1.04)

6. Secondary Outcome: Change From Baseline as Per Investigator's Assessment of Each of the Signs of VVA
Description: Investigator's assessment of vaginal health was performed by visual inspection of the vagina with respect to the signs of VVA: atrophy, pallor, vaginal dryness, friability, and petechiae scored on a 4-point scale where: 0=none, 1=mild, 2=moderate, or 3= severe. The negative change from Baseline indicates improvement. Participants at Final visit/Visit 7 included those who were to complete all the evaluations in the study including who prematurely withdrew from the study.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Previous WC3011 Estradiol Vaginal Cream (2 Times/Week) | Previous Vehicle (2 Times/Week) | Previous WC3011 Estradiol Vaginal Cream (3 Times/Week) | Previous Vehicle (3 Times/Week)
Number analyzed (Participants) | 101 | 56 | 99 | 52
score on a scale
  Atrophy-Baseline | 1.1 (0.70) | 1.5 (0.76) | 1.1 (0.69) | 1.4 (0.80)
  Atrophy-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Atrophy-Change From Baseline to Week 40 | -0.3 (0.79) | -0.7 (0.82) | -0.3 (0.81) | -0.5 (0.77)
  Atrophy-Change From Baseline to Final Visit: number analyzed (Participants) | 97 | 54 | 93 | 48
  Atrophy-Change From Baseline to Final Visit | -0.2 (0.82) | -0.6 (0.80) | -0.2 (0.84) | -0.6 (0.84)
  Pallor-Baseline | 1.1 (0.78) | 1.5 (0.83) | 1.0 (0.74) | 1.3 (0.77)
  Pallor-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Pallor-Change From Baseline to Week 40 | -0.4 (0.81) | -0.8 (1.00) | -0.3 (0.79) | -0.5 (0.77)
  Pallor-Change From Baseline to Final Visit: number analyzed (Participants) | 97 | 54 | 93 | 48
  Pallor-Change From Baseline to Final Visit | -0.4 (0.83) | -0.6 (0.99) | -0.2 (0.82) | -0.6 (0.77)
  Dryness-Baseline | 1.0 (0.81) | 1.4 (0.89) | 1.0 (0.78) | 1.1 (1.01)
  Dryness-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Dryness-Change From Baseline to Week 40 | -0.4 (0.73) | -1.0 (0.92) | -0.4 (0.87) | -0.4 (0.86)
  Dryness-Change From Baseline to Final Visit: number analyzed (Participants) | 97 | 54 | 93 | 48
  Dryness-Change From Baseline to Final Visit | -0.4 (0.75) | -0.8 (0.97) | -0.3 (0.92) | -0.5 (0.94)
  Friability-Baseline | 0.4 (0.67) | 0.6 (0.82) | 0.3 (0.59) | 0.5 (0.75)
  Friability-Change From Baseline to Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Friability-Change From Baseline to Week 40 | -0.2 (0.57) | -0.5 (0.85) | -0.2 (0.67) | -0.2 (0.69)
  Friability-Change From Baseline to Final Visit: number analyzed (Participants) | 97 | 54 | 93 | 48
  Friability-Change From Baseline to Final Visit | -0.2 (0.55) | -0.4 (0.88) | -0.1 (0.73) | -0.3 (0.73)
  Petechiae-Baseline | 0.3 (0.63) | 0.6 (0.80) | 0.2 (0.59) | 0.4 (0.75)
  Petechiae-Change From Baseline at Week 40: number analyzed (Participants) | 84 | 48 | 80 | 42
  Petechiae-Change From Baseline at Week 40 | -0.1 (0.45) | -0.5 (0.80) | -0.1 (0.56) | -0.1 (0.65)
  Petechiae-Change From Baseline to Final Visit: number analyzed (Participants) | 97 | 54 | 93 | 48
  Petechiae-Change From Baseline to Final Visit | -0.1 (0.44) | -0.5 (0.79) | -0.1 (0.54) | -0.2 (0.63)

7. Secondary Outcome: Number of Participants With At Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal (investigational) product, whether or not related to medicinal (investigational) product. TEAE are defined as those AEs with onset date on or after the first dose date of study drug in Study PR-04509, or adverse events that worsen after the first dose date of study drug in Study PR-04509.
Time Frame: Up to Week 40
Population: All participants who received at least 1 dose of study drug in Study PR-04509.
Measure: Count of Participants; unit: Participants
Arm/Group | WC3011 Estradiol Vaginal Cream
Number analyzed (Participants) | 308
Participants | 195

ADVERSE EVENTS:
Time Frame: Up to Week 40
Description: All participants who received at least 1 dose of study drug in Study PR-04509.
Arm/Group | WC3011 Estradiol Vaginal Cream
All-Cause Mortality (participants affected / at risk) | 0/308
Serious Adverse Events (participants affected / at risk) | 8/308
Other Adverse Events (participants affected / at risk) | 50/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WC3011 Estradiol Vaginal Cream (N=308)
Cholelithiasis (Hepatobiliary disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Dysarthria (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Appendicitis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WC3011 Estradiol Vaginal Cream (N=308)
Vulvovaginal Mycotic Infection (Infections and infestations) | 23
Upper Respiratory Tract Infection (Infections and infestations) | 17
Sinusitis (Infections and infestations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.